CLINICAL TRIAL: NCT04992299
Title: Mindfulness-Based Intervention for Depression and Insulin Resistance in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Colorado, Denver (Other); Children's National Research Institute (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-2649; 1U01AT011008 (NIH); 5R01AT011008 (NIH)
Record Dates: First submitted 2021-07-21; First posted 2021-08-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Depression; Insulin Resistance; Obesity; Adolescent Development
Keywords: Adolescent Development; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Insulin Resistance; Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Intervention (Experimental): 6-week group intervention, Learning to BREATHE, an adolescent mindfulness-based intervention derived from mindfulness-based stress reduction
  Interventions: Behavioral: Mindfulness-Based Intervention
- Cognitive-Behavioral Therapy (Active Comparator): 6-week group intervention, the Blues Program, a cognitive-behavioral intervention for adolescents with elevated symptoms of depression
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Health Education (Other): 6-week group program providing didactic information on adolescent health topics
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — 6-week mindfulness-based intervention of 6 weekly 1 hour group sessions
  Arms: Mindfulness-Based Intervention
Behavioral: Cognitive-Behavioral Therapy — 6-week cognitive-behavioral therapy intervention of 6 weekly 1 hour group sessions
  Arms: Cognitive-Behavioral Therapy
Behavioral: Health Education — 6-week health education didactic program of 6 weekly 1 hour group sessions
  Arms: Health Education

SUMMARY:
Rates of type 2 diabetes (T2D) in adolescents have escalated. Adolescent-onset is associated with greater health comorbidities and shorter life expectancy than adult-onset T2D. T2D is preventable by decreasing insulin resistance, a physiological precursor to T2D. T2D prevention standard-of-care is lifestyle intervention to decrease insulin resistance through weight loss; yet, this approach is insufficiently effective in adolescents. Adolescents at risk for T2D frequently experience depression, which predicts worsening insulin resistance and T2D onset, even after accounting for obesity. Mindfulness-based intervention (MBI) may offer a targeted, integrative health approach to decrease depression, and thereby, ameliorate insulin resistance in adolescents at risk for T2D. In a single-site, pilot randomized controlled trial (RCT), we established initial feasibility/acceptability of a 6-week group MBI program, Learning to BREATHE, in adolescents at risk for T2D. We demonstrated feasible single-site recruitment, randomization, retention, protocol adherence, and MBI acceptability/credibility in the target population. Our preliminary data also suggest MBI may lead to greater reductions in stress-related behavior, vs. CBT and a didactic/health education (HealthEd) control group. The current study is multisite, pilot RCT to test multisite fidelity, feasibility, and acceptability in preparation for a future multisite efficacy trial that will have strong external validity, timely recruitment, and long-term follow-up. Adolescents (N=120) at risk for T2D will be randomized to MBI vs. CBT vs. HealthEd and followed for 1-year. Specific aims are to: (1) test multisite fidelity of training and implementation of 6-week group MBI, CBT, and HealthEd, to teens at risk for T2D; (2) evaluate multisite feasibility/acceptability of recruitment, retention, and adherence for an RCT of 6-week group MBI, CBT, HealthEd with 6-week and 1-year follow-up; and (3) modify intervention training/implementation and protocol procedures in preparation for a future, fully-powered multisite efficacy RCT.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent: Age 12-17 years
* At-risk for T2D:

Overweight/obesity: BMI ≥85 percentile for age and sex Family history of T2D: ≥1 relative with T2D, prediabetes, or gestational diabetes in first- or second- degree relative, referring to a biological parent, sibling, aunt, uncle, or grandparent

* Elevated depression symptoms: Center for Epidemiological Studies - Depression Scale (CES-D) total score >20
* Good general health: Medical history/physical examination
* Parent/guardian: Parent/guardian of qualifying participant

Exclusion Criteria:

* Major medical problem: including T2D, assessed at baseline/screening as fasting glucose ≥126 mg/dL or 2-hour glucose ≥200 mg/dL, or any other significant medical condition reported during the medical history/physical examination
* Major psychiatric problem: Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 psychiatric diagnosis, including anorexia nervosa, bipolar disorder, bulimia nervosa, conduct disorder, major depressive disorder (MDD), obsessive compulsive disorder, panic disorder, posttraumatic stress disorder, psychosis, and substance/tobacco/alcohol use disorder
* Regular medication use affecting mood, insulin, and/or weight: anti-anxiety medications, anti-depressants, anti-psychotics, insulin sensitizers, mood stabilizers, stimulants, and weight loss drugs
* Active suicidal ideation or behavior
* Regular psychotherapy or structured weight loss treatment
* Pregnancy: as reported by adolescent participants (females)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Intervention Fidelity | 12-months
  Facilitators score ≥8 on adherence and competence ratings of MBI, CBT, and HealthEd adolescent group sessions (1=poor to 10=exceptional)
Recruitment Feasibility: Percentage of Eligible Adolescents who Enroll | 12-months
  ≥80% eligible adolescents will enroll

SECONDARY OUTCOMES:
Training Fidelity: Facilitator Knowledge after Training | 6-months
  Facilitators score ≥80% on post-training knowledge/ competency tests of MBI, CBT, and HealthEd
Training Fidelity: Facilitator Adherence and Competence during Mock Sessions | 6-months
  Facilitators score ≥8 on adherence and competence ratings of MBI, CBT, and HealthEd mock group sessions (1=poor to 10=exceptional)
Recruitment Feasibility | 12-months
  Attainment of target N=120 within a 12-month period; CONSORT flow/number of months to reach recruitment goal
Intervention Feasibility: Attendance | 6-weeks
  ≥80% adolescents attend 5:6 (80%) group MBI/CBT/HealthEd sessions
Intervention Acceptability: Likeability/Credibility Ratings | 6-weeks
  ≥80% adolescent liking/credibility ratings ≥4 (1=not at all to 5=extremely)
Intervention Acceptability: Qualitative Themes | 6-weeks
  Themes indicative of acceptability of interventions, as derived from grounded theory/qualitative analysis of adolescent focus-groups at post-intervention
Retention Feasibility: Percentage of Adolescents who Complete Follow-ups | 12-months
  ≥80% at post-treatment follow-up and ≥70% at 1-year follow-up
Assessment Feasibility: Percentage Accuracy of Protocols | 18-months
  ≥95% accuracy on standardized protocol checklists for all assessments

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Denver/Children's Hospital Colorado, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Uniformed Services University, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable request.

DOCUMENTS (1):
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT04992299/ICF_001.pdf